CLINICAL TRIAL: NCT01553929
Title: Physical Trainig and Cognitive Activity on the MCI Patient
Brief Title: Physical Training and Cognitive Activity on the Mild Cognitive Impairment (MCI) Patient
Acronym: EPAC-M
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-AOI-03
Record Dates: First submitted 2012-03-08; First posted 2012-03-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: MCI
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Physical and cognitive activity group (Experimental)
  Interventions: Other: Physical Training and cognitive activity (EPC group)
- Physical activity group (Active Comparator)
  Interventions: Other: Physical training (EP group)
- control group (Placebo Comparator)
  Interventions: Other: control group

INTERVENTIONS:
Other: Physical Training and cognitive activity (EPC group) — The patients of the EPC group will realize 2 weekly sessions of 20 minutes of pédalage. During the exercise, the patients will realize a series of tests of decision-making and perceptive cognitive capacity.
  Arms: Physical and cognitive activity group
Other: Physical training (EP group) — The patients of the group (EP) will realize 2 weekly sessions of 20 minutes of pédalage.
  Arms: Physical activity group
Other: control group — no physical training and no cognitive activity
  Arms: control group

SUMMARY:
Regular physical activity is now recognized as a key element of good physical and mental health and this all ages.

MAIN GOAL : Evaluate the effectiveness of physical training associated with a cognitive training in improving the cognitive function of patients diagnosed with Mild Cognitive Impairment (MCI).

DESIGN : Controlled randomized monocentric and prospective study with clinical benefit for the patient with three groups : one physical training and cognitive exercise group, one physical training without cognitive exercise group and one control group.

In agreement with the literature on the effects of physiological stress on cognitive performance, the investigators expect the best cognitive test scores in groups with exercise training compared with controls (35% versus 80% error), and better scores on the MMSE, IALD, depression Scale, Index of Pittsburg sleep quality and quality of Life Questionnaire. Furthermore the investigators hypothesize that this positive effect is greater in the physical training and cognitive exercise group compared with the physical training group only.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patient MCI (Mild Cognitive Impairment)
* Elderly from 40 to 75 years old
* MMSE upper to 22
* Affiliated or beneficiary of a national insurance scheme
* Medical capacity to the physical proposed activity (filling of the conditions of the Medical certificate of not contraindication in the sport)

Exclusion Criteria:

* The placed persons under guardianship, under protection of justice,
* The private persons of freedom (administrative or judicial)
* Nobody already participating in a clinical trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
effectiveness of physical training | up to 3 months
  Assess the effectiveness of physical training associated with a cognitive training in improving the cognitive functions of patients diagnosed with Mild Cognitive Impairment (MCI). We expect the best cognitive test scores in groups with exercise training compared with controls (35% versus 80% error), and better scores on the MMSE, IALD, depression Scale, Index of Pittsburg sleep quality and quality of Life Questionnaire.

SECONDARY OUTCOMES:
Cognitive improvement | up to 3 months
  Assess the cognitive improvement after three months and after cessation of the intervention.
  Assess the impact of the intervention on the cognitive and behavioral, 3 months after cessation of training with maintenance of physical activity by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Franck LE DUFF, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France